CLINICAL TRIAL: NCT05905484
Title: A Phase 1, Double-blind, Single-dose, Randomized, Placebo and Active-Controlled, Four-Way Crossover Study Evaluating the Effects of Bemnifosbuvir on Cardiac Repolarization in Healthy Adult Subjects
Brief Title: Study of Bemnifosbuvir on Cardiac Repolarization in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AT-03A-008
Record Dates: First submitted 2023-04-20; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — AT-511; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Bemnifosbuvir (BEM) therapeutic dose (Experimental): oral tablets
  Interventions: Drug: Bemnifosbuvir (BEM)
- Bemnifosbuvir (BEM) supratherapeutic dose (Experimental): oral tablets
  Interventions: Drug: Bemnifosbuvir (BEM)
- Placebo (Placebo Comparator): oral tablets
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator): oral tablet
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Bemnifosbuvir (BEM) — A single dose of BEM will be administered.
  Other Names: AT-527
  Arms: Bemnifosbuvir (BEM) supratherapeutic dose; Bemnifosbuvir (BEM) therapeutic dose
Drug: Placebo — A single dose of matching placebo will be administered.
  Arms: Placebo
Drug: Moxifloxacin — A single dose of Moxifloxacin will be administered.
  Arms: Moxifloxacin

SUMMARY:
This study will assess the effects of Bemnifosbuvir on cardiac repolarization in healthy Adult Subjects

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug
* Females must have a negative pregnancy test at Screening and prior to dosing
* Minimum body weight of 50 kg and body mass index (BMI) of 18-29 kg/m2
* Willing to comply with the study requirements and to provide written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Infected with hepatitis B virus, hepatitis C virus, HIV or COVID-19
* Abuse of alcohol or drugs
* Use of other investigational drugs within 28 days of dosing
* Other clinically significant medical conditions or laboratory abnormalities

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected (Δ) change-from-baseline QTc (ΔΔQTc). | 24 hours prior to dosing thru 48 hours post dose
  C-QTc analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Québec, Montreal, Quebec, Canada